CLINICAL TRIAL: NCT00490438
Title: Measurement of Vaginal Squeeze Pressure in Incontinent Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Other Study IDs: 06-123
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2006-09

CONDITIONS: Urinary Incontinence
Keywords: perineometry; Modified Oxford Score; pelvic muscles evaluation; urinary incontinence; vaginal palpation
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The patients will be submited to a vaginal squeeze pressure measurements before and after surgeries for urinary incontinence.

DETAILED DESCRIPTION:
Several techniques had been proposed for pelvic floor muscles assessment, however none of them were able to measure the two main functions of these muscles: rising and force of compression. Vaginal palpation is frequently used in clinical evaluation routine and especially the modified Oxford score, but some articles question the Oxford scale sensitivity and its correlation with objective force contraction measurements.

Methods: 45 patients with urinary incontinence treated at the Uroginecology Ambulatory Service of the Hospital de Clínicas de Porto Alegre were included. The patients had been submitted to vaginal palpation using the Oxford score, assessed by a skilled physical therapist, and to the compression force measurement by means of an air filled ballonet connected to a pressure transducer. The two evaluations had been carried in the same day.

ELIGIBILITY:
Inclusion Criteria:

* Stress, urge or mixed stress and urge urinary incontinence.
* Understanding and signing a letter of informed consent

Exclusion Criteria:

* Urinary tract infection.
* Genitourinary surgery during the previous six months.
* Pregnancy or in puerperal period.
* BMI > 40

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-01; Study Completion 2007-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: José G Lopes ramos, Dr, Principal Investigator — Hospital de Clnicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil